CLINICAL TRIAL: NCT03045770
Title: A Randomized, Parallel Control Trial to Compare mFOLFOX Versus mFOLFIRI Versus FOLFPTX (a Combination of Paclitaxel, Fluorouracil) as First-line Treatment in Advanced Gastric Cancer or Adenocarcinoma of Esophagogastric Junction
Brief Title: mFOLFOX Versus mFOLFIRI Versus FOLFPTX as First-line Treatment in AGC or EGJA
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Fujian Cancer Hospital (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FJG201701
Record Dates: First submitted 2017-01-31; First posted 2017-02-07 (Estimated); Last update posted 2017-02-07 (Estimated); Status verified 2017-01

CONDITIONS: Advanced Gastric Cancer Adenocarcinoma of Esophagogastric Junction
MeSH Terms: interventions — Fluorouracil; Oxaliplatin; Irinotecan; Paclitaxel

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- mFOLFOX (Experimental): The mFOLFOX regimen consisted of oxaliplatin (85 mg/m2) and calcium levofolinate (200 mg/m2).Subsequently, a 48-hour infusion of fluorouracil (2400 mg/m2) was administered using an ambulatory pump, repeating the cycle every 14 days till progressive disease or intolerable toxicities.
  Interventions: Drug: Fluorouracil; Drug: Oxaliplatin; Drug: calcium levofolinate
- mFOLFIRI (Experimental): The mFOLFIRI regimen consisted of irinotecan (180 mg/m2) and calcium levofolinate (200 mg/m2).Subsequently, a 48-hour infusion of fluorouracil (2400 mg/m2) was administered using an ambulatory pump, repeating the cycle every 14 days till progressive disease or intolerable toxicities.
  Interventions: Drug: Fluorouracil; Drug: Irinotecan; Drug: calcium levofolinate
- FOLFPTX (Experimental): The FOLFPTX regimen consisted of paclitaxel (95 mg/m2) and calcium levofolinate (200 mg/m2).Subsequently, a 48-hour infusion of fluorouracil (2400 mg/m2) was administered using an ambulatory pump, repeating the cycle every 14 days till progressive disease or intolerable toxicities.
  Interventions: Drug: Fluorouracil; Drug: Paclitaxel; Drug: calcium levofolinate

INTERVENTIONS:
Drug: Fluorouracil — Fluorouracil was used as first line treatment with AGC.
  Other Names: 5-FU
Drug: Oxaliplatin — Oxaliplatin was used as first line treatment with AGC.
  Other Names: OXA
  Arms: mFOLFOX
Drug: Irinotecan — Irinotecan was used as first line treatment with AGC.
  Other Names: CPT-11
  Arms: mFOLFIRI
Drug: Paclitaxel — Paclitaxel was used as first line treatment with AGC.
  Other Names: PTX
  Arms: FOLFPTX
Drug: calcium levofolinate — Calcium levofolinate was used as first line treatment with AGC.

SUMMARY:
The aim of this study was to compare the efficacy and safety of mFOLFOX, mFOLFIRI and FOLFPTX as first-line treatment in AGC or EGJA.

DETAILED DESCRIPTION:
In previous studies, we found that mFOLFOX(a Combination of Oxaliplatin, Fluorouracil), mFOLFIRI(a Combination of Irinotecan, Fluorouracil), FOLFPTX (a Combination of Paclitaxel, Fluorouracil) are active in patients with AGC or EGJA.This study is being done to find out which one has the best efficacy.

ELIGIBILITY:
Inclusion Criteria:

1. Age：18~70years.
2. Subjects with Histologically or cytologically confirmed advanced or metastatic gastric cancer or adenocarcinoma of gastroesophageal junction.
3. First-line treatment patients.
4. subjects with at least one measurable lesion as defined by RECIST (version 1.1).
5. Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1.
6. Survival expectation≥ 3 months.
7. No serious concomitant diseases(including heart,lung,liver jaundice or gastrointestinal obstruction and so on ).
8. Adequate organ functions defined as indicated below： （1）Adequate bone marrow function, defined as: (no blood transfusion within 14 days)

   1. Hemoglobin (Hb)≥80g/L，
   2. White blood count (WBC)≥3.5×109/L
   3. Absolute neutrophil count (ANC)≥1.5×109/L，
   4. Platelet count (PLT)≥75×109/L； （2）Adequate liver function, defined as:

   <!-- -->

   1. Bilirubin ≤1.5×the upper limit of normal (ULN)
   2. Alanine aminotransferase (ALT), or Aspartate aminotransferase (AST) ≤3.0×(ULN), Glutamyl transpeptidase(GGT)≤2.5×(ULN), (When liver metastases, ALT or AST and GPT <5.0×(ULN)).
   3. serum creatinine ≤1.0×（ULN）, or creatinine clearance > 50 mL/min( calculated per the Cockcroft and Gault formula)
9. Females of childbearing potential must be a pregnancy test in 7 days before participating ( including serum or urine), and the results were negative, Females of childbearing potential must agree to use a highly effective method of contraception throughout the entire study period and for 8 weeks after study drug discontinuation. Male subjects must have had a successful vasectomy or they and their female partners must meet the criteria above (i.e.not of childbearing potential or practicing highly effective contraception throughout the study period and for 8 weeks after study drug discontinuation).
10. Subjects provided written informed consent before participating,Willing and able to comply with all aspects of the protocol.

Exclusion Criteria:

1. Females are lactating or pregnant at Screening or Baseline.
2. Patients with other active malignancy (except for definitively treated melanoma in-situ, basal or squamous cell carcinoma of the skin, or carcinoma in-situ of the cervix).
3. Patients who have received previous pre- or post-operative chemotherapy or chemoradiation are ineligible if therapy was completed less than 6 months prior to study registration. Patients must have recovered from adverse events from any previous therapy.
4. Patients with brain or central nervous system metastases, including leptomeningeal disease.
5. Significant cardiac disease as defined as:unstable angina, New York Heart Association (NYHA) grade II or greater, congestive heart failure, history of myocardial infarction within 6 months Evidence of bleeding diathesis or coagulopathy.
6. History of a stroke or CVA within 6 months.
7. Inability to comply with study and/or follow-up procedures.
8. Patients with any other condition that in the opinion of the investigator would preclude his/her participation in a clinical study.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2017-02-10 (Estimated); Primary Completion 2019-12-30 (Estimated); Study Completion 2019-12-30 (Estimated)

PRIMARY OUTCOMES:
Progression-Free Survival (PFS) | 24 months
Adverse Event（AE） | 35 months
  NCI CTC 4.03

SECONDARY OUTCOMES:
Objective Response Rate (ORR) | 24 months
Disease Control Rate (DCR) | 24 months
Overall Survival (OS) | 35 months
Quality of Life (QoL) | 35 months
  Use the validated European Organization for Research and Treatment of Cancer Quality of Life Questionnaire Core 30 [EORTC QLQ-C30].

CONTACTS AND LOCATIONS:
Overall Officials: Jianwei Yang, Principal Investigator — Fujian Cancer Hospital
Locations (1):
- Jianwei Yang, Fuzhou, Fujian, China

IPD SHARING:
Plan to Share IPD: Undecided